CLINICAL TRIAL: NCT06593886
Title: Promoting Upright Mobility in Infants With Cerebral Palsy Using a Robotic Unweighting System
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left NIH
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10001897; 001897-CC
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy; Physical Therapy Modalities; Brain Injuries
Keywords: Mobility; INFANTS; Robotic Unweighting System
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group A (Experimental): This group will participate in active motor training at NIH while using the BabyG device immediately
  Interventions: Device: BabyG
- Group B (Experimental): This group will participate in BabyG training after a 12 week baseline period
  Interventions: Device: BabyG

INTERVENTIONS:
Device: BabyG — This involves wearing a harness connected to the overhead device while in a 10 X 10 play area filled with toys and equipment commonly used for infants to promote mobility skills (e.g. crawling and walking). Families can choose to come for 3 30-minute or 2 45-minute sessions per week. Half of the children will participate in the training immediately after enrollment in the study, the others will wait for 12 weeks before starting training. All will receive a comprehensive assessment at 0, 12 and 24 weeks, with additional developmental assessments at 6 and 18 weeks

SUMMARY:
BabyG is a soft harness attached to a robotic system mounted overhead. While wearing the harness, the infant is free to move around a 10-by-10-foot play area with a padded floor. The harness helps support the infant s weight; it also slows any falls and catches the body before it hits the floor. BabyG can be adjusted to support 5% to 50% of the infant s weight.

Participants will be in the study for 24 weeks, including 12 weeks with BabyG training and 12 weeks without. Training will be 90 minutes per week: either two 45-minute sessions or three 30-minute sessions.

All participants will undergo tests during the 24 weeks such as:

A test to measure an infant s ability to perform tasks such as rolling, sitting, crawling, and walking.

A test to assess nerve function, movements, reflexes, posture, and muscle tone.

A test of brain activity while moving. The infant will be fitted with a snug cap with 64 electrodes. Then the infant will be placed in the BabyG harness and encouraged to take steps on a motorized treadmill. Their movements will be filmed.

DETAILED DESCRIPTION:
Study Description:

This phase IIb randomized crossover trial will evaluate the effects of 12 weeks of mobility training while in a computer-controlled (robotic) unweighting system (BabyG) on motor development rate in infants diagnosed with or at high risk for cerebral palsy (CP) who are less than 18 months old at enrollment compared to a 12-week period when they are not participating in training.

Objectives:

* Primary 1: Evaluate the effects of mobility training with the BabyG robotic unweighting system on motor developmental rate in infants from 5 -18 months compared to an equivalent amount of time when they are not doing the training.
* Primary 2: Evaluate the effects of BabyG mobility training on EEG brain activation patterns during treadmill stepping with the least amount of support needed in infants 5 -18 months, as compared to an equivalent amount of time when they are not doing the training.
* Secondary 1: Evaluate changes in muscle size of the rectus femoris and gastrocnemius muscles as assessed by muscle ultrasound before and after training and compared across training and no-training periods.
* Secondary 2: Relate the age at which the infant starts and their compliance with the BabyG training (total training time) with their

post-training outcomes.

Endpoints:

* Primary Endpoint 1: Compare change in the Bayley IV age equivalents and the GMFM-66 during the training and no-training periods.
* Primary Endpoint 2: Changes in EEG brain activity during supported stepping on an infant treadmill as a result of training. We will quantify and compare changes in the magnitude of activation in multiple EEG frequency bands in motor-related brain regions after

training and no-training periods.

* Secondary Endpoint 1: Changes in brain activation will be correlated w/ changes in Bayley IV and GMFM-66
* Secondary Endpoint 2: The absolute and percent change in muscle size of two muscle groups as a result of training.
* Secondary Endpoint 3: The infant age in months and the total training time in minutes will be correlated with the pre-post change scores on motor, EEG and muscle outcomes

ELIGIBILITY:
* INCLUSION CRITERIA

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. At least 5 months (adjusted for prematurity for those 37 weeks of gestation or less and is based on their due date) and no more than 18 months of age at enrollment
2. A diagnosis of CP or high risk of CP
3. Ability to push up on extended arms in prone for at least 10 seconds or demonstrates an interest in moving from one place to another by rolling, scooting or other means
4. Availability to return to NIH CC with parent or caregiver for training and assessment sessions.

EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Secondary orthopedic, neuromuscular or cardiovascular conditions unrelated to CP that would impede mobility such as hip dysplasia, clubfeet, uncorrected heart defect that affects exertion levels, brachial plexus palsy, among others
2. History of surgery to the upper or lower extremities in the past 6 months
3. Seizure disorder that is not controlled by medication
4. Currently taking baclofen to reduce hypertonia
5. Enrolled in another clinical trial during the study period that involves motor training or other intervention that could influence the outcomes of this study
6. Walk independently for 10 steps on a consistent basis with or without handheld assistive devices.

Ages: 5 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Change in the Bayley IV age equivalents and the GMFM-66 | 48 months
  Compare change in the Bayley IV age equivalents and the GMFM-66 during the training and no-training periods.
Changes in EEG brain activity | 48 months
  Changes in EEG brain activity during supported stepping on an infant treadmill as a result of training. We will quantify and compare changes in the magnitude of activation in multiple EEG frequency bands in motor-related brain regions after training and no-training periods.

SECONDARY OUTCOMES:
Changes in brain activation | 48 months
  Changes in brain activation will be correlated w/ changes in Bayley IV and GMFM-66
The absolute and percent change in muscle size of two muscle groups as a result of training | 48 months
  The absolute and percent change in muscle size of two muscle groups as a result of training
Infant age in months and the total training time in minutes | 48 months
  The infant age in months and the total training time in minutes will be correlated with the pre-post change scores on motor, EEG and muscle outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Damiano, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001897-CC.html